CLINICAL TRIAL: NCT03376828
Title: The Effect of Video and Traditional Laryngoscopy on Hemodynamic Response in Hypertensive and Normotensive Patients
Acronym: Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016/855
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Intubation; Anesthesia; Hypertension
Keywords: laryngoscopy; videolaryngoscopy; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hypertensive T group (Active Comparator): Hypertensive T group: Patients participating in the study were randomly assigned hypertensive (preoperative systolic blood pressure <180 mmHg and diastolic blood pressure <100 mmHg) Macintosh laryngoscopy using intubated
  Interventions: Device: Macintosh laryngoscopy
- Hypertensive VL group (Active Comparator): Hypertensive VL group: Patients participating in the study were randomly assigned hypertensive (preoperative systolic blood pressure <180 mmHg and diastolic blood pressure <100 mmHg) C-Mac Videolaryngoscope using intubated
  Interventions: Device: C-Mac Videolaryngoscope
- Non-hypertensive T group (Sham Comparator): Non-hypertensive T group: (Preoperative systolic blood pressure < 140 mmHg and diastolic blood pressure < 100 mmHg) Macintosh laryngoscopy using intubated
  Interventions: Device: Macintosh laryngoscopy
- Non-hypertensive VL group (Sham Comparator): Non-hypertensive VL group: Preoperative systolic blood pressure < 140 mmHg and diastolic blood pressure < 100 mmHg C-Mac Videolaryngoscope using intubated
  Interventions: Device: C-Mac Videolaryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscopy — Endotracheal intubation time using the Macintosh laryngoscope
  Arms: Hypertensive T group; Non-hypertensive T group
Device: C-Mac Videolaryngoscope — Endotracheal intubation time using the C-Mac Videolaryngoscope
  Arms: Hypertensive VL group; Non-hypertensive VL group

SUMMARY:
During endotracheal intubation, it is known that la laryngoscopy has significant effects, such as tachycardia and blood pressure increase, which may be harmful, especially in those with cardiovascular disease. Different studies comparing laryngeal stimulation and there resulting hemodynamic response made with various intubation devices are available in the literature. The investigators planned to work with the hypothesis that endotracheal intubation with videolaryngoscopy would have less hemodynamic response traditional (Macintosh) laryngoscopy and the use of videolaryngoscopy would result in wider vision with less laryngeal stimulation.

DETAILED DESCRIPTION:
In this study, in a study on endotracheal intubation under general anesthesia, a routine preparation of endotracheal intubation using video laryngoscopy or Macintosh laryngoscopy in adult hypertensive and normotensive patients between 18-75 years old, form will be written and recorded.

Patient age, weight, height, sex, operation, co-morbid conditions and vital findings, measurements used in airway evaluation, initial trial success, laryngoscope using number of procedures, intubation tube number will be recorded.

Statistical analysis was performed using statistical program to compare the hemodynamic response of hypertensive and normotensive patients using videolaryngoscope or Macintosh laryngoscope

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years.
* Underwent surgery under general anesthesia.

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) IV, V patients
* Preoperative systolic blood pressure 180 mmHg, diastolic blood pressure a pressure above 110 mmHg.
* Ejection fraction is less than 40%.
* Difficult intubation history
* Mallampati 3,4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Hemodynamic response | 0-10 minute
  Change from baseline noninvasive blood pressure and heart rate

SECONDARY OUTCOMES:
intubation time | 0-120 seconds
  The time elapsed between the passage of the laryngoscopy through the teeth to teeth
Glottic view grade | During intubation
  Using the Cormack Lehane score

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)

REFERENCES:
- [Background] Kihara S, Brimacombe J, Yaguchi Y, Watanabe S, Taguchi N, Komatsuzaki T. Hemodynamic responses among three tracheal intubation devices in normotensive and hypertensive patients. Anesth Analg. 2003 Mar;96(3):890-895. doi: 10.1213/01.ANE.0000048706.15720.C9. PMID 12598280
- [Background] Abdelgawad AF, Shi QF, Halawa MA, Wu ZL, Wu ZY, Chen XD, Yao SL. Comparison of cardiac output and hemodynamic responses of intubation among different videolaryngoscopies in normotensive and hypertensive patients. J Huazhong Univ Sci Technolog Med Sci. 2015 Jun;35(3):432-438. doi: 10.1007/s11596-015-1449-7. Epub 2015 Jun 14. PMID 26072085
- [Background] Sarkilar G, Sargin M, Saritas TB, Borazan H, Gok F, Kilicaslan A, Otelcioglu S. Hemodynamic responses to endotracheal intubation performed with video and direct laryngoscopy in patients scheduled for major cardiac surgery. Int J Clin Exp Med. 2015 Jul 15;8(7):11477-83. eCollection 2015. PMID 26379966
- [Background] McCoy EP, Mirakhur RK, McCloskey BV. A comparison of the stress response to laryngoscopy. The Macintosh versus the McCoy blade. Anaesthesia. 1995 Nov;50(11):943-6. doi: 10.1111/j.1365-2044.1995.tb05924.x. PMID 8678248
- [Background] Hossfeld B, Frey K, Doerges V, Lampl L, Helm M. Improvement in glottic visualisation by using the C-MAC PM video laryngoscope as a first-line device for out-of-hospital emergency tracheal intubation: An observational study. Eur J Anaesthesiol. 2015 Jun;32(6):425-31. doi: 10.1097/EJA.0000000000000249. PMID 25886716